CLINICAL TRIAL: NCT05549245
Title: RCT Study of Short-term Clinical Efficacy of High Flow Nasal Catheter Oxygen Therapy for Obstructive Sleep Apnea
Brief Title: Clinical Efficacy of High-flow Nasal Cannula Oxygen Therapy in Patients With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022038
Record Dates: First submitted 2022-08-14; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Continues Positive Airway Pressure; High-flow Nasal Cannula Oxygen Therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow Nasal Cannula Oxygen Therapy group (Experimental)
  Interventions: Device: high-flow nasal cannula oxygen therapy,
- Continues Positive Airway Pressure group (Other)
  Interventions: Device: CPAP

INTERVENTIONS:
Device: high-flow nasal cannula oxygen therapy, — Patients were treated with high-flow nasal cannula oxygen therapy for three nights
  Arms: High-flow Nasal Cannula Oxygen Therapy group
Device: CPAP — Patients were treated with CPAP for three nights
  Arms: Continues Positive Airway Pressure group

SUMMARY:
Patients meeting the criteria of obstructive sleep apnea were included, and all patients signed informed consent, which met the requirements of the ethics Committee of our unit. All subjects were hospitalized patients. Subjects were randomly enrolled into High-flow Nasal Cannula Oxygen Therapy group or Continues Positive Airway Pressure group for 3 days of treatment. Sleep monitoring was performed on the first and fourth day of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. There were typical symptoms of sleep snoring at night with apnea and daytime sleepiness (ESS score ≥9). Stenosis and obstruction in any part of the upper airway were observed on physical examination, with AHI≥5 times /h.
2. For patients with no significant daytime sleepiness (ESS score < 9), AHI≥10 times /h.
3. Patients with AHI≥5 times /h had one or more OSAHS complications, such as cognitive impairment, hypertension, coronary heart disease, cerebrovascular disease, diabetes and insomnia.

Exclusion Criteria:

1. Patients who cannot tolerate non-invasive ventilator or transnasal high-flow oxygen therapy.
2. Ongoing treatment may affect sleep, such as sedatives, hypnotics, muscle relaxants, etc.
3. Hemodynamic instability.
4. Severe respiratory diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
AHI | The first day of enrollment
  Apnea Hypopnea Index:The number of episodes of sleep apnea per hour
AHI | The fourth day of enrollment
  Apnea Hypopnea Index:The number of episodes of sleep apnea per hour
Treatment failure rate | The fourth day of enrollment
  Number of patients unable to tolerate treatment/enrollment
Good compliance rate | The fourth day of enrollment
  Number of patients treated for more than 4 hours per night/enrolled
longest apnea time | The first day of enrollment
  Maximum duration(s) of nocturnal sleep apnea in patients
longest apnea time | The fourth day of enrollment
  Maximum duration(s) of nocturnal sleep apnea in patients
Mean oxygen saturation | The first day of enrollment
  Mean oxygen saturation during the patient's night sleep
Mean oxygen saturation | The fourth day of enrollment
  Mean oxygen saturation during the patient's night sleep
minimum oxygen saturation | The first day of enrollment
  Lowest oxygen saturation during the patient's night sleep
minimum oxygen saturation | The fourth day of enrollment
  Lowest oxygen saturation during the patient's night sleep

SECONDARY OUTCOMES:
Gender | The first day of enrollment
  Male and female
height | The first day of enrollment
  Height (in cm)
age | The first day of enrollment
  years
weight | The first day of enrollment
  Kg
total sleep time | The first day of enrollment
  Total sleep duration(min) of the patient at night
total sleep time | The fourth day of enrollment
  Total sleep duration(min) of the patient at night
Number of awakening | The first day of enrollment
  The number of awakenings during the patient's night sleep
Number of awakening | The fourth day of enrollment
  The number of awakenings during the patient's night sleep

CONTACTS AND LOCATIONS:
Overall Officials: enqi Zhao, master, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordan AS, McSharry DG, Malhotra A. Adult obstructive sleep apnoea. Lancet. 2014 Feb 22;383(9918):736-47. doi: 10.1016/S0140-6736(13)60734-5. Epub 2013 Aug 2. PMID 23910433
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Background] Parke RL, McGuinness SP. Pressures delivered by nasal high flow oxygen during all phases of the respiratory cycle. Respir Care. 2013 Oct;58(10):1621-4. doi: 10.4187/respcare.02358. Epub 2013 Mar 19. PMID 23513246
- [Background] Nakanishi N, Suzuki Y, Ishihara M, Ueno Y, Tane N, Tsunano Y, Itagaki T, Oto J. Effect of High-Flow Nasal Cannula on Sleep-disordered Breathing and Sleep Quality in Patients With Acute Stroke. Cureus. 2020 Jul 20;12(7):e9303. doi: 10.7759/cureus.9303. PMID 32832300
- [Background] Yan H, Qinghua L, Mengyuan P, Yaoyu C, Long Z, Mengjie L, Xiaosong D, Fang H. High flow nasal cannula therapy for obstructive sleep apnea in adults. Sleep Breath. 2022 Jun;26(2):783-791. doi: 10.1007/s11325-021-02453-6. Epub 2021 Aug 12. PMID 34383275
- [Background] Nilius G, Wessendorf T, Maurer J, Stoohs R, Patil SP, Schubert N, Schneider H. Predictors for treating obstructive sleep apnea with an open nasal cannula system (transnasal insufflation). Chest. 2010 Mar;137(3):521-8. doi: 10.1378/chest.09-0357. Epub 2009 Dec 1. PMID 19952061